CLINICAL TRIAL: NCT06180226
Title: Evaluation of Brain Functional Changes With 18F-FDG PET and Cognitive Processes After Brain Radiotherapy for Cavernous Sinus Meningiomas and Non-secreting ACTH Adenomas
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: MENINGIOMA/RADIOTOSS
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET CT with 18 FDG . — Impact exerted by the use of 18FDG PET in the process of functional monitoring of the patient undergoing radiotherapy treatment.

SUMMARY:
The use of radiotherapy for irradiation of all or part of the brain, in the treatment of extracerebral intracranial neoplasms, is growing rapidly, both due to the increase in diagnoses of primary tumors thanks to new imaging methods, and for the increase in the number of new cases of cancer.

Cerebral neurotoxicity linked to radiation treatment is an adverse effect that is not always accurately evaluated based on the prognosis of some brain pathologies. The progression of diagnostic and therapeutic methods has recently generated a modification of therapeutic protocols and some categories of radiotreated patients may incur acute, subacute and late effects. These include manifestations of acute neurological deterioration, more frequently effects classified as sub-acute such as "somnolence syndrome" (from 2 to 6 weeks after the end of treatment) and finally late effects, which manifest themselves as a variety of neurological deficits in particular a decline in cognitive brain functions, probably linked to a direct effect on neurons or the result of an imbalance in the connections between white matter and cerebral gray matter. In relation to the myelin function of conduction of axonal transmission, the result of radio-induced damage in this site would manifest itself with a significant reduction in the speed of transmission of the impulse and consequently with a dramatic worsening of cognitive processes. In particular, clinically, radiologically and in some cases also from a pathological point of view, the damage from rays on the brain parenchyma would have aspects similar to those of a degenerative pathology such as Alzheimer's disease. These effects are usually measured on the patient by subjective assessments or using neuropsychological tests. The use, not only experimental, of neurophysiological methods for the study of cognitive processes in neurology and in degenerative disorders such as dementia is increasingly frequent. These methods are based on the study of specific neuronal circuits involved in the cognitive functions of the human brain in normal conditions and in the presence of pathology. Among the techniques that allow an analysis of molecular alterations in vivo there are scintigraphic ones, i.e. nuclear medicine ones, including single photon emission tomography (SPET) and positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* lesion dimensions compatible with a GAmma Knife treatment or tomotherapy;
* adequate hematological, hepatic and renal function;
* signed informed consent.

Exclusion Criteria:

* patients < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting with a cyto/histological diagnosis of cavernous sinus meningioma or intracranial and extracerebral neoplasia.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-04-21 (Actual); Primary Completion 2014-12-11 (Actual); Study Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
PET CT with 18 FDG in adult patients affected by extracerebral intracranial cavernous sinus meningioma. | 6 years
  evaluation of the impact of the use of 18 FDG PET in the process of functional monitoring of patients undergoing radiotherapy treatment.

IPD SHARING:
Plan to Share IPD: No